CLINICAL TRIAL: NCT05010382
Title: Efficacy of Two Dental Implants With Different Surface Characteristics in Patients With History of Periodontitis. A Randomized Controlled Clinical Trial.
Brief Title: Efficacy of Implant Surface Characteristics in Patients With History of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Ti Care S.L (Unknown)
Responsible Party: Principal Investigator, Benjamín Serrano Torrecilla, Doctorate student, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17.516-R_P
Record Dates: First submitted 2021-08-03; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Marginal Bone Loss
Keywords: Implant surface; hybrid; Peri-implantitis; Periodontitis; Marginal bone loss
MeSH Terms: conditions — Peri-Implantitis; Periodontitis

STUDY DESIGN:
Intervention Model Description: Patients will recieve an implant with either hybrid surface (test group) or moderately rough surface (control implants
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Hybrid surface dental implant
  Interventions: Procedure: Implant placement surgery
- Control group (Experimental): moderately rough surface implant
  Interventions: Procedure: Implant placement surgery

INTERVENTIONS:
Procedure: Implant placement surgery — Under local anaesthesia, full-thickness mucoperiosteal flaps were elevated, the alveolar ridge measured, and a proper implant dimension (3.75 mm and 4.25 mm diameter; 8 mm, 10 mm and 11.5 mm length) and position selected. After site preparation, each patient was randomly allocated to the test or the control group. Patients in the test group received a modified implant design with the coronal third presenting a machined surface (hybrid surface (HS) group), while in the control group the same implant design with a titanium rough surface up to the implant shoulder was used (rough surface (RS) group). Implants were placed 1 mm sub-crestally. In the case of dehiscence or fenestrations around the implant, the patient was excluded from the study. Once inserted, healing abutments (ranging between 3 -5 mm) were placed, and flaps sutured around the abutments to allow for a transmucosal healing.

SUMMARY:
The aim of the study is to evaluate in patients with history of periodontitis the clinical, microbiological and radiological outcomes of implants with a modified implant design consisting on a machined surface in the coronal third of the implant.

In this 12-month, parallel-arm, randomized controlled trial, patients with history of treated periodontitis and in need of dental implants for single-unit or short edentulous spaces (i.e. two implants) will be randomly assigned to a test group (implants with a hybrid surface, presenting a machined coronal third; HS) or a control group (conventional moderately rough implants; RS). Implants will be restored 3 months later with fixed implant supported reconstructions. Radiological, clinical, microbiological and patient-related outcome measures (PROMs) will be assessed 3, 6 and 12 months after the prosthetic installation.

ELIGIBILITY:
Inclusion Criteria:

•> 20 years of age

* Presence of ≥1 adjacent missing teeth, in either maxilla or mandible (up to three missing units).
* A natural tooth had to be present mesially to the most proximal implant site, although free end situations were allowed, and opposing dentition had to be natural teeth or implant supported fixed restorations.
* History of treated and controlled periodontitis.
* Presence of adequate bone volume to achieve primary implant stability without concomitant regeneration

Exclusion Criteria:

* Diseases affecting bone metabolism or wound healing (e.g.)
* History of radiation therapy, leukocyte dysfunction, or any other immunodeficiency
* Drug abuse
* Intrasurgical exclusion criteria, such as the lack of primary stability, the need of bone augmentation or the impossibility of placing the implant based on prosthetic requirements. �

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
Radiographic marginal bone levels Change | Change between baseline and 12 months
  Radiographic marginal bone levels (bone loss) are defined as the distance between the bone crest and the implant shoulder at mesial and distal sites.
  For standardization of periapical radiographs the same film holder-beam aiming device will be applied (Rinn System) and silicone custom-made bite blocks will be used to improve reproducible repositioning. All digital radiographs will be evaluated by one calibrated and trained researcher (BS) using a software (AutoCAD® Autodesk ®, California, USA) that allows to calibrate the distances using the known implant length.

SECONDARY OUTCOMES:
Clinical periodontal outcome measurements change | Change between baseline and 12 months
  Clinical measurements will be performed at six sites per implant of i) probing depth (PD), ii) marginal mucosa recession assessed as length of the implant crown (CLI; distance from the mucosal margin to the oclusal surface at the mid buccal point), iii) bleeding on probing (BoP) and iv) plaque scores (PI). Finally, peri-implant mucositis, defined as the presence of profuse BoP.
Microbiologic outcome measurements change | Change between baseline and 12 months
  Paper points will be inserted to the depth of the peri-implant pocket and kept in place for 15 sec. The points will be transferred into a screw-capped vial, containing 1.5 ml of reduced transport fluid, (RTF) and maintained at -20ºC. Microbiological analysis by means of anaerobic culture will be performed for the determination of counts, proportion and frequency of detection of Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Prevotella intermedia and Fusobacterium nucleatum.�
Patient reported outcome measures (PROM's)change | Change between baseline and 12 months
  PROM´s will be assessed by means of a questionnaire comprising 4 items: comfort, appearance, masticatory function and overall satisfaction. Patients will be asked to rate these four aspects according to the following scale: very unsatisfied, unsatisfied, fair, satisfied and very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz Alonso, Chair, Study Chair — Universidad Complutense de Madrid
Locations (1):
- Facultad de odontología, Complutense University of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buser D, Sennerby L, De Bruyn H. Modern implant dentistry based on osseointegration: 50 years of progress, current trends and open questions. Periodontol 2000. 2017 Feb;73(1):7-21. doi: 10.1111/prd.12185. PMID 28000280
- [Background] Cochran DL. A comparison of endosseous dental implant surfaces. J Periodontol. 1999 Dec;70(12):1523-39. doi: 10.1902/jop.1999.70.12.1523. PMID 10632528
- [Background] Polizzi G, Gualini F, Friberg B. A two-center retrospective analysis of long-term clinical and radiologic data of TiUnite and turned implants placed in the same mouth. Int J Prosthodont. 2013 Jul-Aug;26(4):350-8. doi: 10.11607/ijp.3386. PMID 23837166
- [Background] John G, Becker J, Schwarz F. Modified implant surface with slower and less initial biofilm formation. Clin Implant Dent Relat Res. 2015 Jun;17(3):461-8. doi: 10.1111/cid.12140. Epub 2013 Aug 27. PMID 23981274
- [Background] Teughels W, Van Assche N, Sliepen I, Quirynen M. Effect of material characteristics and/or surface topography on biofilm development. Clin Oral Implants Res. 2006 Oct;17 Suppl 2:68-81. doi: 10.1111/j.1600-0501.2006.01353.x. PMID 16968383
- [Background] Esposito M, Murray-Curtis L, Grusovin MG, Coulthard P, Worthington HV. Interventions for replacing missing teeth: different types of dental implants. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD003815. doi: 10.1002/14651858.CD003815.pub3. PMID 17943800
- [Background] Albouy JP, Abrahamsson I, Berglundh T. Spontaneous progression of experimental peri-implantitis at implants with different surface characteristics: an experimental study in dogs. J Clin Periodontol. 2012 Feb;39(2):182-7. doi: 10.1111/j.1600-051X.2011.01820.x. Epub 2011 Dec 4. PMID 22136592
- [Background] Albouy JP, Abrahamsson I, Persson LG, Berglundh T. Spontaneous progression of peri-implantitis at different types of implants. An experimental study in dogs. I: clinical and radiographic observations. Clin Oral Implants Res. 2008 Oct;19(10):997-1002. doi: 10.1111/j.1600-0501.2008.01589.x. PMID 18828815
- [Background] Albouy JP, Abrahamsson I, Persson LG, Berglundh T. Implant surface characteristics influence the outcome of treatment of peri-implantitis: an experimental study in dogs. J Clin Periodontol. 2011 Jan;38(1):58-64. doi: 10.1111/j.1600-051X.2010.01631.x. Epub 2010 Nov 24. PMID 21092053
- [Background] Donati M, Ekestubbe A, Lindhe J, Wennstrom JL. Marginal bone loss at implants with different surface characteristics - A 20-year follow-up of a randomized controlled clinical trial. Clin Oral Implants Res. 2018 May;29(5):480-487. doi: 10.1111/clr.13145. Epub 2018 Mar 23. PMID 29569767
- [Background] Wennstrom JL, Ekestubbe A, Grondahl K, Karlsson S, Lindhe J. Oral rehabilitation with implant-supported fixed partial dentures in periodontitis-susceptible subjects. A 5-year prospective study. J Clin Periodontol. 2004 Sep;31(9):713-24. doi: 10.1111/j.1600-051X.2004.00568.x. PMID 15312092
- [Background] Aglietta M, Siciliano VI, Rasperini G, Cafiero C, Lang NP, Salvi GE. A 10-year retrospective analysis of marginal bone-level changes around implants in periodontally healthy and periodontally compromised tobacco smokers. Clin Oral Implants Res. 2011 Jan;22(1):47-53. doi: 10.1111/j.1600-0501.2010.01977.x. Epub 2010 Sep 10. PMID 20831754
- [Background] Hinode D, Tanabe S, Yokoyama M, Fujisawa K, Yamauchi E, Miyamoto Y. Influence of smoking on osseointegrated implant failure: a meta-analysis. Clin Oral Implants Res. 2006 Aug;17(4):473-8. doi: 10.1111/j.1600-0501.2005.01244.x. PMID 16907781
- [Background] Roccuzzo M, Bonino F, Aglietta M, Dalmasso P. Ten-year results of a three arms prospective cohort study on implants in periodontally compromised patients. Part 2: clinical results. Clin Oral Implants Res. 2012 Apr;23(4):389-95. doi: 10.1111/j.1600-0501.2011.02309.x. Epub 2011 Sep 28. PMID 22092445
- [Background] Matarasso S, Rasperini G, Iorio Siciliano V, Salvi GE, Lang NP, Aglietta M. A 10-year retrospective analysis of radiographic bone-level changes of implants supporting single-unit crowns in periodontally compromised vs. periodontally healthy patients. Clin Oral Implants Res. 2010 Sep;21(9):898-903. doi: 10.1111/j.1600-0501.2010.01945.x. Epub 2010 Apr 20. PMID 20438576
- [Background] Karoussis IK, Salvi GE, Heitz-Mayfield LJ, Bragger U, Hammerle CH, Lang NP. Long-term implant prognosis in patients with and without a history of chronic periodontitis: a 10-year prospective cohort study of the ITI Dental Implant System. Clin Oral Implants Res. 2003 Jun;14(3):329-39. doi: 10.1034/j.1600-0501.000.00934.x. PMID 12755783
- [Background] Gallego L, Sicilia A, Sicilia P, Mallo C, Cuesta S, Sanz M. A retrospective study on the crestal bone loss associated with different implant surfaces in chronic periodontitis patients under maintenance. Clin Oral Implants Res. 2018 Jun;29(6):557-567. doi: 10.1111/clr.13153. Epub 2018 Apr 17. PMID 29664148
- [Background] Zetterqvist L, Feldman S, Rotter B, Vincenzi G, Wennstrom JL, Chierico A, Stach RM, Kenealy JN. A prospective, multicenter, randomized-controlled 5-year study of hybrid and fully etched implants for the incidence of peri-implantitis. J Periodontol. 2010 Apr;81(4):493-501. doi: 10.1902/jop.2009.090492. PMID 20367092
- [Background] Pikner SS, Grondahl K, Jemt T, Friberg B. Marginal bone loss at implants: a retrospective, long-term follow-up of turned Branemark System implants. Clin Implant Dent Relat Res. 2009 Mar;11(1):11-23. doi: 10.1111/j.1708-8208.2008.00092.x. Epub 2008 Apr 1. PMID 18384403
- [Derived] Serrano B, Sanz-Sanchez I, Montero E, Sanz M. Three-Year Outcomes of Dental Implants With a Hybrid Surface Macro-Design Placed in Patients With History of Periodontitis: A Randomised Clinical Trial. J Clin Periodontol. 2025 Jun;52(6):802-812. doi: 10.1111/jcpe.14153. Epub 2025 Apr 25. PMID 40277088
- [Derived] Serrano B, Sanz-Sanchez I, Serrano K, Montero E, Sanz M. One-year outcomes of dental implants with a hybrid surface macro-design placed in patients with history of periodontitis: A randomized clinical trial. J Clin Periodontol. 2022 Feb;49(2):90-100. doi: 10.1111/jcpe.13575. Epub 2021 Dec 14. PMID 34881442